CLINICAL TRIAL: NCT00465413
Title: Bronchodilatation Effects of a Small Volume Spacer Used With a Metered-Dose Inhaler
Acronym: MDI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMH-I-S-317
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-09

CONDITIONS: Asthma
Keywords: metered-dose inhalers (MDI); forced expiratory volume in 1 second (FEV1); forced expiratory flow rate (FEF25-75%)
MeSH Terms: conditions — Asthma | interventions — Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Small volume spacer and/or Rinsing the mouth with water

SUMMARY:
The purpose of the present study is to determine whether use of a small volume spacer is associated with better bronchodilatation in an unselected population of patients with documented reversible airflow limitations.

DETAILED DESCRIPTION:
Administration of bronchodilator drugs with metered-dose inhalers (MDIs) is difficult for some patients because the timing of the spray and the inhalation must be coordinated exactly. Use of spacers seems to improve delivery in these patients. It is not clear, however, if there is any advantage to a spacer for patients who are able to use an MDI with correct technique.

The purpose of the present study is to determine whether use of a small volume spacer is associated with better bronchodilatation in an unselected population of patients with documented reversible airflow limitations. The intervention in the first part of the study is use of an MDI with or without a spacer to deliver a bronchodilator (2 puffs, 0.4 mg of fenoterol). Spirometry is performed before and after the inhalation.

The second part of the study is conducted identically to the first with the same conditions and variables but with the addition of rinsing the mouth with 100 mL of water after inhaling the bronchodilator but before the second spirometry measurement.

The outcome to be measured is the increase in forced expiratory volume in 1 second (FEV1) and forced expiratory flow rate (FEF25-75%).

ELIGIBILITY:
Inclusion Criteria:

* age > 6 years old,
* subjects known to have reversible airway limitation with demonstrated response to bronchodilators on spirometry.

Exclusion Criteria:

* refusal to participate,
* negative bronchodilator test,
* poor performance of pulmonary function testing.

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-09

PRIMARY OUTCOMES:
forced expiratory volume in 1 second (FEV1)
forced expiratory flow rate (FEF25-75%)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Lung Liu, MD, Study Chair — Mackay Memorial Taitung Branch Hospital; Yen-Ta Lu, MD, PhD., Principal Investigator — Mackay Memorial Tamshui Branch Hospital
Locations (2):
- Taiwan (2):
  - Mackay Memorial Tamshui Branch Hospital, Tamshui, Taipei
  - Mackay Memorial Taitung Branch Hospital, Taitung, Taitung

REFERENCES:
- [Derived] Liu CL, Lu YT. Bronchodilatation effects of a small volume spacer used with a metered-dose inhaler. J Asthma. 2009 Sep;46(7):637-41. doi: 10.1080/02770900802492111. PMID 19728196
- See also: Home page of Mackay Memorial Hospital — http://www.mmh.org.tw/